CLINICAL TRIAL: NCT01147614
Title: Brief CBT for Pediatric Anxiety and Depression in Primary Care
Brief Title: Brief Cognitive Behavioral Therapy (CBT) for Pediatric Anxiety and Depression in Primary Care
Acronym: BCBT-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of Pittsburgh (Other); Kaiser Permanente (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, V. Robin Weersing, Associate Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7887933; 5R01MH084935 (NIH)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Anxiety; Depression
Keywords: Child; adolescent; anxiety; depression; internalizing; cognitive behavioral therapy; pediatric primary care
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- specialty mental health care referral (Active Comparator)
  Interventions: Behavioral: Specialty mental health care referral (SMHC)
- Brief Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy (BCBT)

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy (BCBT) — BCBT: 8-12 sessions over 16 weeks of cognitive-behavioral therapy administered by Master's-level clinicians in primary care setting
  Other Names: BCBT
  Arms: Brief Cognitive Behavioral Therapy
Behavioral: Specialty mental health care referral (SMHC) — SMHC: specialty mental health care referrals provided
  Other Names: SMHC
  Arms: specialty mental health care referral

SUMMARY:
The purpose of this study is to determine whether a brief (12 week) psychological treatment program, based in primary care, can help youths struggling with anxiety and/or depression. This brief cognitive behavioral therapy program will be compared to enhanced referral to specialty mental health care.

DETAILED DESCRIPTION:
Mood and anxiety disorders in childhood and adolescence are disabling, distressing, and prevalent and produce added costs to health systems. This two-site randomized controlled trial will test the effects of a brief cognitive behavioral therapy (BCBT) protocol (8-12 sessions) in a large sample (N=210) of children and adolescents (age 8-16) presenting with anxiety and/or depression in primary care. Clinical and cost-effectiveness of BCBT will be compared to a plausible public health alternative - enhanced referral to specialty mental health care (SMHC). This investigation is noteworthy in adopting a deployment-focused model and testing this intervention early in its development within a real world context (primary care) and against a plausible public health comparison condition (SMHC) relevant for future treatment dissemination.

ELIGIBILITY:
Inclusion Criteria:

* meet full or probable diagnostic criteria for Separation Anxiety Disorder, Generalized Anxiety Disorder, Social Phobia, Major Depression, Dysthymic Disorder, or Minor Depression
* age 8.0 to 16.9
* live with legal, consenting guardian for at least 6 months

Exclusion Criteria:

* youths requiring alternate intervention (e.g., youths with bipolar disorder, psychosis, active suicidal ideation with plan, PTSD, substance dependence, current physical or sexual abuse, or mental retardation
* suffer from serious or unstable physical illness (e.g., uncontrolled diabetes)
* currently in active, alternate intervention for anxiety or depression (e.g., antidepressant use)

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2010-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression | measured at baseline (week 0)
Clinical Global Impression | measured at post-treatment (week 16)
Clinical Global Impression | measured at 8 month follow-up (week 32)

SECONDARY OUTCOMES:
Pediatric Anxiety Rating Scale | measured at baseline (week 0)
Children's Depression Rating Scale - Revised | measured at baseline (week 0)
Health Utilities Index | measured at baseline (week 0)
  This measure will aid in cost-effectiveness analyses.
Pediatric Anxiety Rating Scale | measured at post-treatment (week 16)
Pediatric Anxiety Rating Scale | measured at 8 month follow-up (week 32)
Children's Depression Rating Scale - Revised | measured at post-treatment (week 16)
Children's Depression Rating Scale - Revised | measured at 8 month follow-up (week 32)
Health Utilities Index | measured at post-treatment (week 16)
  This measure will aid in cost-effectiveness analyses.
Health Utilities Index | measured at 8 month follow-up (week 32)
  This measure will aid in cost-effectiveness analyses.

CONTACTS AND LOCATIONS:
Overall Officials: V. Robin Weersing, Ph.D., Principal Investigator — San Diego State University; David A Brent, M.D., Principal Investigator — Western Psychiatric Institute and Clinics
Locations (2):
- United States (2):
  - San Diego State University, San Diego, California
  - Western Psychiatric Institute and Clinics, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Weersing VR, Gonzalez A, Campo JV, Lucas AN. Brief behavioral therapy for pediatric anxiety and depression: Piloting an integrated treatment approach. Cognitive and Behavioral Practice 15: 126-139, 2008.
- [Derived] Baca SA, Goger P, Glaser D, Rozenman M, Gonzalez A, Dickerson JF, Lynch FL, Porta G, Brent DA, Weersing VR. Reduction in avoidance mediates effects of brief behavioral therapy for pediatric anxiety and depression. Behav Res Ther. 2023 May;164:104290. doi: 10.1016/j.brat.2023.104290. Epub 2023 Mar 8. PMID 36965232
- [Derived] Schwartz KTG, Kado-Walton M, Dickerson JF, Rozenman M, Brent DA, Porta G, Lynch FL, Gonzalez A, Weersing VR. Brief Behavioral Therapy for Anxiety and Depression in Pediatric Primary Care: Breadth of Intervention Impact. J Am Acad Child Adolesc Psychiatry. 2023 Feb;62(2):230-243. doi: 10.1016/j.jaac.2022.08.007. Epub 2022 Aug 24. PMID 36030033
- [Derived] Brent DA, Porta G, Rozenman MS, Gonzalez A, Schwartz KTG, Lynch FL, Dickerson JF, Iyengar S, Weersing VR. Brief Behavioral Therapy for Pediatric Anxiety and Depression in Primary Care: A Follow-up. J Am Acad Child Adolesc Psychiatry. 2020 Jul;59(7):856-867. doi: 10.1016/j.jaac.2019.06.009. Epub 2019 Jul 3. PMID 31278996
- [Derived] Weersing VR, Brent DA, Rozenman MS, Gonzalez A, Jeffreys M, Dickerson JF, Lynch FL, Porta G, Iyengar S. Brief Behavioral Therapy for Pediatric Anxiety and Depression in Primary Care: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jun 1;74(6):571-578. doi: 10.1001/jamapsychiatry.2017.0429. PMID 28423145
- See also: Click here for more information about this study: Brief CBT for Pediatric Anxiety and Depression in Primary Care — http://www.sci.sdsu.edu/chaamp/
- See also: Click here for more information about this study: Brief CBT for Pediatric Anxiety and Depression in Primary Care — http://www.Pedspittnet.pitt.edu